CLINICAL TRIAL: NCT00363272
Title: A PHASE 1 STUDY OF ISPINESIB (SB-715992) IN PEDIATRIC PATIENTS WITH RELAPSED OR REFRACTORY SOLID TUMORS
Brief Title: Ispinesib in Treating Young Patients With Relapsed or Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01828; ADVL0517; U01CA097452 (NIH); CDR0000491407 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Burkitt Lymphoma; Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Spinal Cord Neoplasm; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Burkitt Lymphoma; Choroid Plexus Neoplasms; Astrocytoma; Spinal Cord Neoplasms; Familial ependymoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma | interventions — ispinesib; CK0238273

ARMS (1):
- Arm I (Experimental): Patients receive ispinesib IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of ispinesib in treating young patients with relapsed or refractory solid tumors or lymphoma. Drugs used in chemotherapy, such as ispinesib, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of ispinesib in pediatric patients with refractory solid tumors or lymphoma.

II. Define and describe the toxicities of ispinesib in these patients. III. Characterize the pharmacokinetics of ispinesib in these patients.

SECONDARY OBJECTIVES:

I. Define, preliminarily, the antitumor activity of ispinesib. II. Determine the relationship between CYP3A4 gene polymorphisms and pharmacokinetics in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive ispinesib IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ispinesib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients undergo blood and tumor sample collection periodically for pharmacokinetic and gene polymorphism correlative studies.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy at either original diagnosis or relapse, including the following:

  * Solid tumor, including primary CNS tumors

    * Neurologic deficits in patients with CNS tumors must have been relatively stable for ≥ 1 week
    * Patients with CNS tumors must be on stable or decreasing doses of dexamethasone for the past 7 days
    * Histology requirement waived for intrinsic brain stem tumors
  * Lymphoma
* Measurable or evaluable disease
* No known curative therapy or no therapy proven to prolong survival with an acceptable quality of life exists
* Patients with known bone marrow metastases are eligible for study but are not evaluable for hematologic toxicity

  * Not known to be refractory to red blood cell or platelet transfusions
* Karnofsky performance score (PS) 60-100% (> 10 years of age) or Lansky PS 60-100% (≤ 10 years of age)
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to study enrollment)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine based on age as follows:

  * No greater than 0.8 mg/dL (≤ 5 years of age)
  * No greater than 1.0 mg/dL (6 to 10 years of age)
  * No greater than 1.2 mg/dL (11 to 15 years of age)
  * No greater than 1.5 mg/dL (> 15 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal
* ALT ≤ 45 U/L
* Albumin ≥ 2 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of active graft-vs-host disease
* No uncontrolled infection
* Recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* More than 1 week since prior growth factors, including those that support platelet or WBC number or function
* At least 1 week since prior biologic agents
* At least 2 weeks since prior local, palliative, small-port external-beam radiotherapy
* At least 6 months since prior total body irradiation (TBI), craniospinal radiotherapy, or radiotherapy to ≥ 50%of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy (i.e., skull, spine, pelvis, or ribs)
* At least 3 months since prior stem cell transplantation or rescue without TBI
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No concurrent enzyme-inducing anticonvulsants, including any of the following:

  * Phenytoin
  * Phenobarbital
  * Felbamate
  * Primdone
  * Oxcarbazepine
  * Carbamazepine
* No concurrent agents that inhibit CYP3A4, including any of the following:

  * Itraconazole
  * Ketoconazole
  * Voriconazole

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the maximum dose at which fewer than one-third of patients experience DLT, graded according to NCI CTCAE version 3.0 | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sills, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States